CLINICAL TRIAL: NCT03955770
Title: Effects of High Flow Oxygen Therapy on Exercise Performance in Patients With Chronic Obstructive Pulmonary Disease. A Randomized, Controlled Trial.
Brief Title: Effects of HFOT on Exercise Performance in Patients With COPD. A Randomized, Controlled Trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01-8/464-15
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Exercise endurance; High-flow oxygen therapy; Low-flow oxygen therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFOT first then LFOT (Experimental)
  Interventions: Combination Product: High-flow oxygen therapy (HFOT); Combination Product: Low-flow oxygen therapy (LFOT)
- LFOT first then HFOT (Experimental)
  Interventions: Combination Product: High-flow oxygen therapy (HFOT); Combination Product: Low-flow oxygen therapy (LFOT)

INTERVENTIONS:
Combination Product: High-flow oxygen therapy (HFOT) — HFOT will be applied by a dedicated large bore nasal cannula (Optiflow+, Fisher&Paykel, New Zealand) at a flow rate 60 L/min, FiO2 45%, temperature 32 °C, using a HFOT device (myAIRVO2, Fisher&Paykel, New Zealand).
Combination Product: Low-flow oxygen therapy (LFOT) — LFOT will be provided by a standard nasal cannula at a flow rate of 3 L/min using an oxygen concentrator (EverFlow, Philips Respironics).

SUMMARY:
This will be a randomized, cross-over trial evaluating the efficacy of nasal high-flow oxygen therapy (HFOT) vs. low-flow oxygen therapy (LFOT) on cycling endurance in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This will be a randomized, cross-over trial evaluating the efficacy of nasal HFOT vs. LFOT on cycling endurance in patients with COPD. Each patient will perform two constant load cycling exercise tests to exhaustion using HFOT and LFOT on two consecutive days, respectively, according to randomization. The load of the cycle ergometer will be set at 75% of the individually estimated maximum work rate (Wmax). During exercise tests, LFOT will be provided by a standard nasal cannula at a flow rate of 3 L/min using an oxygen concentrator. HFOT will be applied by a dedicated large bore nasal cannula at a flow rate 60 L/min, FiO2 45%, temperature 32 °C, using a HFOT device.

ELIGIBILITY:
Inclusion criteria:

Men and women, 35 to 75 years of age, with moderate to severe COPD, (FEV1/FVC <0.7, FEV1 40-80% predicted, resting SpO2 ≥92%, PaCO2 <6 kPa at 760 m) who live <800 m will be invited.

Exclusion criteria:

COPD exacerbation, very severe COPD with hypoxemia (FEV1/FVC <0.7, FEV1 <40% predicted, oxygen saturation on room air <92%), current heavy smoking (>20 cigarettes per day), comorbidities such as uncontrolled cardiovascular disease, internal, neurologic, rheumatologic or psychiatric disease that interfere with protocol compliance.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Exercise endurance time in seconds | HFOT on day 1 vs. LFOT on day 2 or vice versa, according to randomization
  Difference in the exercise endurance time between HFOT vs. LFOT during a constant load exercise test at 75% of the maximal work capacity.

SECONDARY OUTCOMES:
Dyspnea sensation | HFOT on day 1 vs. LFOT on day 2 or vice versa, according to randomization
  Difference in the exercise induced dyspnea sensation between HFOT vs LFOT assessed by the BORG CR10 scale ranging from 0 "no dyspnea at all" to 10 "Maximum of dyspnea" assessed at the end of exercise.
Subjective leg fatigue sensation | HFOT on day 1 vs. LFOT on day 2 or vice versa, according to randomization
  Difference in the exercise induced subjective leg fatigue sensation between HFOT vs LFOT assessed by the BORG CR10 scale ranging from 0 "no leg fatigue at all" to 10 "Maximum of leg fatigue" assessed at the end of exercise.
Arterial blood gases | HFOT on day 1 vs. LFOT on day 2 or vice versa, according to randomization
  Difference of parameters in the arterial blood gases, in particular pH, SaO2, PaO2 and PaCO2 between HFOT vs. LFOT at the end of exercise.
Heart rate in bpm | HFOT on day 1 vs. LFOT on day 2 or vice versa, according to randomization
  Difference in the maximal heart rate assessed by ECG between HFOT vs. LFOT at the end of exercise.
Arterial blood pressure in mmHg | HFOT on day 1 vs. LFOT on day 2 or vice versa, according to randomization
  Difference in the maximal blood pressure between HFOT vs. LFOT at the end of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Furian, PhD, Principal Investigator — University Hospital, Zürich; Konrad E Bloch, MD, Study Chair — University of Zurich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

REFERENCES:
- [Derived] Bitos K, Furian M, Mayer L, Schneider SR, Buenzli S, Mademilov MZ, Sheraliev UU, Marazhapov NH, Abdraeva AK, Aidaralieva SD, Muratbekova AM, Sooronbaev TM, Ulrich S, Bloch KE. Effect of High-Flow Oxygen on Exercise Performance in COPD Patients. Randomized Trial. Front Med (Lausanne). 2021 Feb 19;7:595450. doi: 10.3389/fmed.2020.595450. eCollection 2020. PMID 33693009